CLINICAL TRIAL: NCT02104791
Title: Procalcitonin Has a Role to Play in Prediction of Intra-amniotic Subclinical Infection.
Brief Title: Evaluation of the Role of Plasma Procalcitonin in Prediction of Intra-amniotic Infection in Preterm Premature Rupture of Membrane
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Alaa Sayed Hassanin, Lecturer, Ain Shams Maternity Hospital
Other Study IDs: MRCOG-1988
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Intra-amniotic Subclinical Infection.
Keywords: Procalcitonin; intra-amniotic subclinical infection.
MeSH Terms: interventions — Procalcitonin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- procalcitonin in blood: -Group 1: Healthy preterm Group: will include 50 pregnant females all at 24-34 weeks of gestational age .
  Interventions: Drug: procalcitonin
- plasma of blood: -Group 2: Preterm premature rupture of membrane Group include 50 pregnant women
  Interventions: Drug: procalcitonin
- procalcitonin,prematureruptureofmembrane in blood: Complete history including (special habits like smoking and alcohol taking, menstrual history especially LMP, medical diseases, past obstetric history including duration, mode of delivery for each pregnancy, and if there were fetal or maternal complications).
  Physical examination including (general condition, height, weight, vital signs).-Ultrasound to execlude multiple pregnancies, IUFD and to confirm oligohydraminos in group2.
  The venous blood samples will be taken for measuring of -Procalcitonin in mothors -CRP and WBCs in mothers to detect infection -CRP in neonates of mothers of group 2.
  They will be asked for their permission and consent.
  Interventions: Drug: procalcitonin

INTERVENTIONS:
Drug: procalcitonin — In patient with preterm premature rupture of membrane (PPROM) is the procalcitonin can be used to predict intra-amniotic subclinical infection?
  Other Names: plasma

SUMMARY:
It is hypothesized that the procalcitonin has a role to play in prediction of intra-amniotic subclinical infection.

DETAILED DESCRIPTION:
Study population

* This study will be conducted at the department of Obstetrics and Gynecology recruiting pregnant women selected from the attendees of antenatal clinic, emergency department and from inpatient wards of Ain Shams University Maternity Hospital from Mars2014.
* This study will include 100 pregnant women these cases will be divided into 2 groups:
* Group 1: Healthy preterm Group: will include 50 pregnant females all at 24-34 weeks of gestational age .
* Group 2: Preterm premature rupture of membrane Group: will include 50 pregnant females all at 24-34 weeks of gestational age

ELIGIBILITY:
Patients are with singleton pregnancies. Rupture of membranes will be diagnosed by history, sterile speculum examination to confirm fluid leakage from the cervical canal and ultrasound to confirm oligohydraminos.

Subclinical infection will be detected with laboratory indices (WBC count of ≥15, 000 c/mm3, CRP of ≥1 mg/dL) without any clinical symptoms and signs of infection as urinary tract infection in group 1 patients.

Women with multiple pregnancies. Clinical signs of infection as (fever,abdominal tendernes). Cervical dilatations of 2 cm or more. Maternal disease like diabetes or fetal complications like intra-uterine fetal death.

Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population
  * This study will be conducted at the department of Obstetrics and Gynecology recruiting pregnant women selected from the attendees of antenatal clinic, emergency department and from inpatient wards of Ain Shams University Maternity Hospital from Mars2014.
  * This study will include 100 pregnant women these cases will be divided into 2 groups:
  * Group 1: Healthy preterm Group: will include 50 pregnant females all at 24-34 weeks of gestational age .
  * Group 2: Preterm premature rupture of membrane Group: will include 50 pregnant females all at 24-34 weeks of gestational age.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
The correlation between procalcitonin level in PPROM and C-reactive protein level in neonates. | one year
  The correlation between procalcitonin level in PPROM and C-reactive protein level in neonates

SECONDARY OUTCOMES:
Procalcitonin. - C-reactive protein. - White blood cells count (total and diffrantiated). -C-reactive protein in neonates of groub 2. | one year
  Procalcitonin.
  * C-reactive protein.
  * White blood cells count (total and diffrantiated).
  * C-reactive protein in neonates of groub 2.

OTHER OUTCOMES:
Procalcitonin. - C-reactive protein. - White blood cells count (total and diffrantiated). -C-reactive protein in neonates of groub 2. | one year
  Procalcitonin.
  * C-reactive protein.
  * White blood cells count (total and diffrantiated).
  * C-reactive protein in neonates of groub 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Result] Oludag T, Gode F, Caglayan E, Saatli B, Okyay RE, Altunyurt S. Value of maternal procalcitonin levels for predicting subclinical intra-amniotic infection in preterm premature rupture of membranes. J Obstet Gynaecol Res. 2014 Apr;40(4):954-60. doi: 10.1111/jog.12273. Epub 2013 Dec 10. PMID 24320627